CLINICAL TRIAL: NCT06689228
Title: Principal Investigator
Brief Title: The Effect of Education Based on Orem's Self-Care Deficit Theory and Tele-Monitoring on Rational Drug Use in Haemodialysis Patients
Acronym: Haemodialysis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hatice CEYLAN, Asisstant Professor, Akdeniz University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/197; Hatice CEYLAN (Registry Identifier: The Effect of Web Based Education Based on Self-Care Deficiency Theory on Self-Care Power and Self-Efficacy and Perceiv)
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Haemodialysis
Keywords: haemodialysis; Orem; Rational Drug use; Nurses

STUDY DESIGN:
Intervention Model Description: Orem's Self-Care Deficit Theory and Tele-Monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Randomized (Experimental): The Effect of Education Based on Self-Care Deficiency Theory on Rational Drug Use in Patients Receiving Haemodialysis In the study, which will last for 2 months, the patients in the intervention group will receive pre-test training based on the Self-Care Deficiency Theory. Also weekly reminder messages will be sent regularly.
  Other Names:
  Education Based on Self-Care Deficiency Theory on Rational Drug Use
  Interventions: Other: Rational Drug Use Training

INTERVENTIONS:
Other: Rational Drug Use Training — Rational Drug Use Training and Tele-monitoring will include information on drugs and their importance, rational drug use, rational drug use in haemodialysis patients, harms of irrational drug use, benefits of rational drug use, obstacles encountered in rational drug use, ways to overcome obstacles encountered in rational drug use, and increasing self-efficacy. The first training is planned to last approximately 30-35 minutes for each patient and the second training (summary training) is planned to last approximately 15-20 minutes. With telemonitoring, reminder messages will be sent to patients' phones at intervals.
  Other Names: Tele-monitoring

SUMMARY:
Patients with chronic kidney disease may show altered pharmacokinetic and pharmacodynamic response to many drugs compared to patients with normal renal function. Therefore, effective and safe drug use is difficult in patients with chronic kidney disease and especially in dialysis patients. In addition, some drugs may have nephrotoxic effects by causing further deterioration in renal function, especially in high-risk renal patients. Prevention of problems related to drug use in haemodialysis patients will be possible with rational drug use (RUD). RDM is defined as 'the set of rules to be followed in order for patients to take medicines in accordance with their clinical needs, in doses that meet their personal needs, in sufficient time, at the lowest cost to themselves and the society'.

Rational drug use has become an increasingly important concept today. In studies investigating rational drug use, problems such as incorrect use of drugs, prescribing more drugs than necessary, unnecessary injection recommendation/administration, unnecessary antibiotic consumption, and unnecessary use of expensive drugs have been identified. As a result of incorrect drug use, poisoning or decreased sensitivity to drugs are observed.

DETAILED DESCRIPTION:
The Effect of Education Based on Orem's Self-Care Deficit Theory and Tele-Monitoring on Rational Drug Use in Haemodialysis Patients

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* No communication or medically recognised mental problems,
* Patients receiving haemodialysis treatment for 6 months or longer were included in the study.

Exclusion Criteria:

* Diagnosed with psychiatric illness
* Diagnosed with malignancy
* Individuals who do not allow access to their information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Rationanl Drug use Scale | two months
  The Rational Drug Use Scale (RUDS) consists of 21 items and one dimension (Appendix 3). The items are scored on a 5-point Likert-type scale (1-Never, 2-Rarely, 3-Sometimes, 4-Most of the time and 5-Always) according to their fulfilment of the statements. Only the 17th item in the scale is reversed. After the reversed item is reversed, the sum of all scale items gives the 'total scale score'. The total score of the EHRS varies between 21 and 105. As the total score obtained from AİKÖ increases, rational drug use increases. When evaluating the total score obtained from AİKÖ; if the total score obtained is between 21- 52, it is scored as low level, between 53-67 as medium level, and between 68-105 as high level.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided